CLINICAL TRIAL: NCT07192887
Title: Clinical Feasibility of Thebaine Urine Mass Spectrometry Drug Testing
Brief Title: Thebaine Urine Testing
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0818
Record Dates: First submitted 2025-06-12; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Urine Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To develop and validate a urine drug screen to detect thebaine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Ages 18-65
* Healthy

Exclusion Criteria:

* Allergy to poppy seeds, or any of the related food stuffs used in the study
* Celiac disease or gluten sensitivity
* Ongoing or opioid use in the past 6 months
* History of renal or hepatic disease or dysfunction
* Inability or unwillingness to give repeated urine specimens
* Unwillingness to refrain from eating poppy seed-containing products during the two-day course of the study
* Non-English speakers (due to study materials being in English)
* BMI greater than 30
* Antibiotic use in the previous 2 months
* Recent ingestion of poppy seeds from the previous 7 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Flyers will be posted throughout the medical center for recruiting.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Validate thebaine urine screen | Enrollment to 48 hours after enrollment
  Validate a liquid chromatography-tandem mass spectrometry method to detect thebaine in urine

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Walter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No